CLINICAL TRIAL: NCT07154303
Title: Smartphone-Based Use of Phonocardiography, Electrocardiography Accessory, and/or Facial Photoplethysmography to Detect Atrial Fibrillation: Diagnostic Performance Study
Brief Title: Testing the Performance of Smartphones and Their Accessories in Detecting Irregularly Irregular Heart Rhythm
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Laboratory of Data Discovery for Health (Unknown)
Responsible Party: Principal Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: AUSC/ECG/rPPG-AF; UW 24-763 (Other: Institutional Review Board of The University of Hong Kong/Hospital Authority Hong Kong West Cluster)
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Smartphone; Persistent Atrial Fibrillation; Mobile Health; mHealth; Telemedicine; Artificial Intelligence; Heart Sounds; Phonocardiography; Photoplethysmography; Electrocardiography; 12-Lead ECG; 12-Lead EKG; 12-Lead Electrocardiography; ECG; EKG; Electrocardiogram; Electrocardiograph
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial Fibrillation
  Interventions: Diagnostic Test: Computer algorithms
- Sinus Rhythm
  Interventions: Diagnostic Test: Computer algorithms

INTERVENTIONS:
Diagnostic Test: Computer algorithms — Computer algorithms that are designed to perform heart sound, electrocardiography (ECG), and/or facial photoplethysmography (rPPG) analysis on data collected from smartphone's internal hardware and/or external accessories.
  Other Names: ausculto®; Vitogram®; FacialAI

SUMMARY:
The purpose of this 4-in-1 observational study is to test the performance of artificial intelligences (AIs) in distinguishing irregularly irregular heart rhythm called atrial fibrillation (AF) from normal heart rhythm using physiological signals collected by smartphones' built-in hardware and/or external accessories.

Participants will:

* Have their weight, height, resting heart rate and blood pressures measured
* Have 12-lead electrocardiogram (ECG) of their heart electrical activities recorded
* Have their heart sounds and 1-lead ECG recorded from their chest, and optical-based blood flow data (photoplethysmography or PPG) and 1-lead ECG recorded from their fingers using smartphones' built-in microphone, camera, and/or external accessories
* Optionally have their optical-based blood flow data recorded from their face using smartphones' built-in camera (remote PPG or rPPG).

The researchers will also create a database containing the physiological signals collected in this study along with the participants' medically relevant information to help train and test future AIs for medical applications.

DETAILED DESCRIPTION:
4 observational studies have been combined into 1 observational study to share the same pool of participants. These 4 studies are designated as AUSC-AF, ECG-AF, AUSC+ECG-AF, and rPPG-AF corresponding to the signal modality/modalities used for AF detection (see outcome measures) and designated as AUSC/ECG/rPPG-AF when combined as 1 study.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥22 years (adult)
* Patients who have one of the following:
* Permanent atrial fibrillation, or
* Long-standing persistent atrial fibrillation (12 months or longer), or
* Confirmed 12-lead ECG diagnosis for persistent atrial fibrillation (> 7 days) or sinus rhythm within 12 months at the time of their normal attendance at the hospital

Exclusion Criteria:

Any of the following:

* Implanted active medical devices in the torso, such as pacemakers and defibrillators
* Patients without atrial fibrillation who have another arrhythmia
* Completely missing one or more limbs, or missing any hand
* Disability in using their hands or arms
* Lack of both index fingers, or all fingers in any hand
* Both index fingers with any of the following characteristics:
* Tattooed/inked
* Reduced blood flow in the fingertip (e.g. perniosis or callus formation)

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospital cardiology patients
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Differentiation of Atrial Fibrillation from Sinus Rhythm in Heart Sound Recordings | Day 0
  AUSC-AF: Identification of atrial fibrillation (AF) from sinus rhythm in recorded heart sounds (phonocardiogram [PCG]) as verified by the gold standard 12-lead electrocardiography (ECG) interpretation, measured in the form of sensitivity and specificity.

SECONDARY OUTCOMES:
Differentiation of Atrial Fibrillation from Sinus Rhythm in Heart Sound Recordings | Day 0
  AUSC-AF: Identification of atrial fibrillation from sinus rhythm in recorded heart sounds (phonocardiogram [PCG]) as verified by the gold standard 12-lead ECG interpretation, measured in the form of positive and negative predictive values, and accuracy.
Differentiation of Atrial Fibrillation from Sinus Rhythm in 1-Lead ECG Signals | Day 0
  ECG-AF: Identification of atrial fibrillation from sinus rhythm in recorded 1-lead ECG signals as verified by the gold standard 12-lead ECG interpretation, measured in the form of sensitivity, specificity, positive and negative predictive values, and accuracy.
Differentiation of Atrial Fibrillation from Sinus Rhythm in PCG and 1-Lead ECG Signals | Day 0
  AUSC+ECG-AF: Identification of atrial fibrillation from sinus rhythm in PCG and 1-lead ECG signals as verified by the gold standard 12-lead ECG interpretation, measured in the form of sensitivity, specificity, positive and negative predictive values, and accuracy.
Differentiation of Atrial Fibrillation from Sinus Rhythm in Facial Photoplethysmography Signals | Day 0
  rPPG-AF: Identification of atrial fibrillation from sinus rhythm in facial photoplethysmography signals (also known as remote photoplethysmography [rPPG]) as verified by the gold standard 12-lead ECG interpretation, measured in the form of sensitivity, specificity, positive and negative predictive values, and accuracy.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No